CLINICAL TRIAL: NCT04117763
Title: Effect of EMPAgliflozin on The HeterogeneitY of Ventricular Repolarization in Patients With Diabetes and Coronary HEART Disease.
Brief Title: Effect of Empagliflozin on Ventricular Repolarization.
Acronym: EMPATHYHEART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Caramelli, Associated Professor of Medicine, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 99613518.9.0000.0068
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Heart Disease; Arrythmia, Cardiac
Keywords: empagliflozin; Diabetes; coronary heart disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Disease; Arrhythmias, Cardiac; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Patient data will be compared before and after treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Experimental): Empagliflozin 25 mg once daily for 3 months
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Empagliflozin once daily, for three months

SUMMARY:
The present project aims to investigate if the empagliflozin has an antiarrhythmic action. Analyzing the T-wave heterogeneity index, a new electrocardiographic risk marker associated with the prediction of cardiovascular risk, in diabetic patients and coronary artery disease, the investigators will verify if empagliflozin is associated with a reduction in electrical instability.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of morbidity and mortality in diabetic patients.

New hypoglycemic drugs are required to undergo cardiovascular safety studies for their release. In 2015, EMPA-REG OUTCOME, which was done for empagliflozin´s approval was the first study to provide evidence that an antidiabetic agent could decrease cardiovascular events. The results demonstrated a reduction in the primary outcome (death by cardiovascular causes, nonfatal infarction, and nonfatal stroke), cardiovascular mortality and hospitalization for heart failure in patients with type 2 diabetes at high cardiovascular risk who received empagliflozin in combination with standard treatment. It is noteworthy that the study population was under-optimized clinical treatment with antihypertensives, statin and aspirin and especially it is noteworthy that the difference in the primary outcome over placebo became evident only three months after treatment´s start.

The potential mechanisms underlying the surprising cardiovascular benefits of empagliflozin are not fully understood.

The present project aims to investigate if the empagliflozin has an antiarrhythmic action. Analyzing the T-wave heterogeneity index, a new electrocardiographic risk marker associated with the prediction of cardiovascular risk, in diabetic patients and coronary artery disease, we will verify if empagliflozin is associated with a reduction in electrical instability.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years;

  * Fasting glycemia> 100 mg/dl or previous diagnosis of type 2 diabetes mellitus;
  * Coronary artery disease, defined by one of the following criteria: the antecedent of myocardial infarction; the evidence of significant coronary stenosis in previous coronary angiography; the noninvasive positive test for ischemia (stress electrocardiogram, stress echocardiogram, stress scintigraphy)
  * TWH ≥ 80 microvolts

Exclusion Criteria:

* Chronic renal insufficiency with glomerular filtration rate ≤ 45 ml / min / 1.73m2;
* Hepatic insufficiency (determined by Child-Pugh, B or C classification);
* Age ≥ 85 years;
* 12-lead resting electrocardiogram with the following changes: intraventricular conduction disorders (bundle branch block), pacemaker rhythm, atrial fibrillation or flutter, artifact stroke distortion or baseline fluctuation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Arrhythmogenic burden | 3 months
  Analysis of the T-wave heterogeneity index

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Caramelli, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- InCor, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No